CLINICAL TRIAL: NCT04924036
Title: A Prospective Trial to Assess How Glycopyrronium Cloths at the Amputation Site of Limb Amputees Changes the Severity of Hyperhidrosis and the Fit and Function of the Prosthetic Measured by Patient Reported Outcomes
Brief Title: Qbrexza Cloths for Hyperhidrosis of Amputation Sites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Stephanie Z Klein, Assistant Professor, Dermatology, Principal Investigator, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00139912
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Amputation; Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Intervention Model Description: This is a Prospective, Double Blinded, Placebo Controlled, Randomized, Cross-over trial.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators in the trial will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Glycopyrronium Cloths then Placebo (Other): Participants that are randomized to Glycopyrronium cloths for 4 weeks, then 2 week wash out, then cross over to placebo cloths for 4 weeks.
  Interventions: Drug: glycopyrronium cloths; Drug: Placebo
- Placebo then Glycopyrronium Cloths (Other): Participants that are randomized to placebo cloths for 4 weeks, then 2 week wash out, then cross over to Glycopyrronium cloths for 4 weeks.
  Interventions: Drug: glycopyrronium cloths; Drug: Placebo

INTERVENTIONS:
Drug: glycopyrronium cloths — Qbrexza is an anticholinergic indicated for topical treatment of axillary hyperhidrosis in adults and pediatric patients 9 years of age and older
  Other Names: Qbrexza Cloths
Drug: Placebo — Placebo for this study are cloths that look like the qbrexza cloths but do not have any active ingredient.

SUMMARY:
This is a Prospective, Double Blinded, Placebo Controlled, Randomized, Cross-over trial using Qbrexza Cloths to treat hyperhidrosis of amputation sites. There is a 2 week screening period where patients will use an activity monitor to establish baseline activity level, then patients will be randomized to receive either Qbrexza cloths or placebo for 4 weeks, then a 2 week washout, and then a 4-week cross-over treatment period.

DETAILED DESCRIPTION:
BACKGROUND:

Approximately 1 in 190 people in the United States have experienced a limb amputation. Of these patients with amputations, over sixty percent suffer from hyperhidrosis at the amputation site. Amputation site hyperhidrosis interferes with these patients' daily activities as well as their ability to engage in vigorous activity beneficial to their overall health. In fact, amputees identified heat and sweating as what reduces their quality of life more than any other problem, even pain. Despite the significant impact hyperhidrosis has on amputees' quality of life and ability to stay physically active, there are no self-administered, non-invasive, well-tolerated treatments for amputation site hyperhidrosis. Botulinum toxin injections are an available treatment option for focal hyperhidrosis. However, the large surface area covered by the prosthetic and prosthetic sleeve often necessitates very large volumes of botulinum toxin for effective treatment at amputation sites. This is costly, making it difficult to be able to treat the entire affected area. Botulinum toxin also requires office visits and repeat treatments every 4-6 months.

Glycopyrronium cloths are a unique treatment possibility, because they can easily be used over a large body surface area and can easily be self-administered at home. At this time, glycopyrronium cloths are only FDA approved for use in the axillae. There are two primary differences between the use of these cloths at amputation sites and axillae: 1) the amputation site is occluded during daytime hours by the prosthetic and 2) the area treated for amputation-site hyperhidrosis (the entire area covered by the prosthetic sleeve) is typically a much larger surface area than the axillae. These factors could significantly increase systemic absorption of glycopyrronium and cause systemic side effects. In order to minimize these effects, the medication will be applied at night, when the site is not occluded. Frequent visits with the investigator will also encourage early reporting of symptoms which could be the result of systemic side effects associated with use on a larger surface area. Patient reported outcomes will be used to determine effectiveness.

This is a Prospective, Double Blinded, Placebo Controlled, Randomized, Cross-over trial.

Participants will be randomized, using a 1:1 ratio, to one of 2 arms:

* Arm #1: At Baseline participants will receive active treatment for 4 weeks, completing a 1 week wash out period and then concluding with 4 weeks of placebo treatment
* Arm #2: At baseline participants will receive placebo for 4 weeks, completing a 1 week washout period and then concluding with active treatment for 4 weeks.

Primary Objective 1. Determine if daily use of glycopyrronium cloths applied to the amputation site decreases hyperhidrosis severity and improved fit and function of the prosthetic as measured by patient reported outcome measures.

Primary Endpoints

1. Determine the change in ASDD-m Impact scores between the end of the treatment and placebo periods.

ELIGIBILITY:
Inclusion Criteria:

1. History of limb amputation with limb-amputation surgery at least 6 months ago
2. Have a prosthetic device

4. HDSS of 3 or greater (at screening) 5. ASDD-m Item 2 severity score >= 4 (at screening) 6. PFFQ score >= 4 (at screening)

Exclusion Criteria:

1. Open sores or wounds on residual limb (at screening and baseline)
2. Known sensitivity to glycopyrronium tosylate or other component of Qbrexza
3. Pregnant or lactating.
4. Use of botulinum toxin within 1 year of the baseline visit
5. Use of topical aluminum chloride within 1 month of the baseline visit
6. Any significant concurrent condition that could adversely affect the patient's participation and/or the assessment of the safety and efficacy in the study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2023-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Z Klein, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah MidValley Dermatology, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chren MM. The Skindex instruments to measure the effects of skin disease on quality of life. Dermatol Clin. 2012 Apr;30(2):231-6, xiii. doi: 10.1016/j.det.2011.11.003. Epub 2011 Dec 20. PMID 22284137
- [Background] Hagberg K, Branemark R. Consequences of non-vascular trans-femoral amputation: a survey of quality of life, prosthetic use and problems. Prosthet Orthot Int. 2001 Dec;25(3):186-94. doi: 10.1080/03093640108726601. PMID 11860092
- [Background] Hansen C, Godfrey B, Wixom J, McFadden M. Incidence, severity, and impact of hyperhidrosis in people with lower-limb amputation. J Rehabil Res Dev. 2015;52(1):31-40. doi: 10.1682/JRRD.2014.04.0108. PMID 26230919
- [Background] Strutton DR, Kowalski JW, Glaser DA, Stang PE. US prevalence of hyperhidrosis and impact on individuals with axillary hyperhidrosis: results from a national survey. J Am Acad Dermatol. 2004 Aug;51(2):241-8. doi: 10.1016/j.jaad.2003.12.040. PMID 15280843
- [Background] Nelson LM, DiBenedetti D, Pariser DM, Glaser DA, Hebert AA, Hofland H, Drew J, Ingolia D, Gillard KK, Fehnel S. Development and validation of the Axillary Sweating Daily Diary: a patient-reported outcome measure to assess axillary sweating severity. J Patient Rep Outcomes. 2019 Sep 5;3(1):59. doi: 10.1186/s41687-019-0148-8. PMID 31486951
- [Background] Lamb YN. Topical Glycopyrronium Tosylate in Primary Axillary Hyperhidrosis: A Profile of Its Use. Clin Drug Investig. 2019 Nov;39(11):1141-1147. doi: 10.1007/s40261-019-00853-x. PMID 31571127
- [Background] Solish N, Bertucci V, Dansereau A, Hong HC, Lynde C, Lupin M, Smith KC, Storwick G; Canadian Hyperhidrosis Advisory Committee. A comprehensive approach to the recognition, diagnosis, and severity-based treatment of focal hyperhidrosis: recommendations of the Canadian Hyperhidrosis Advisory Committee. Dermatol Surg. 2007 Aug;33(8):908-23. doi: 10.1111/j.1524-4725.2007.33192.x. PMID 17661933
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618

RESULTS

PARTICIPANT FLOW:
Groups:
- Glycopyrronium Cloths, Then Placebo: Participants Randomized Glycopyrronium Cloths, then Placebo.
  Participants first received glycopyronium cloths for 4 weeks, then a 1 week washout period, and then 4 weeks of placebo.
  glycopyrronium cloths: Qbrexza is an anticholinergic indicated for topical treatment of axillary hyperhidrosis in adults and pediatric patients 9 years of age and older
- Placebo, Then Glycopyrronium Cloths: Participants were randomized to placebo cloths for 4 weeks, then a 1-week washout period, and then 4 weeks with the glycopyrronium cloths.
  Placebo: Placebo for this study are cloths that look like the glycopyrronium cloths but do not have any active ingredient.
Period: Overall Study
Arm/Group | Glycopyrronium Cloths, Then Placebo | Placebo, Then Glycopyrronium Cloths
Started | 7 | 6
Completed | 3 | 4
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycopyrronium Cloths Then Placebo | Placebo Then Glycopyrronium Cloths | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (14.9) | 43.6 (14.1) | 43.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: ASDD-m Sweat Severity Score
Description: ASDD-m is a questionnaire for axillary hyperhidrosis measuring for presence, severity, impact and bothersomeness of the patient's sweating. Question #1 is "Rate the Sweating at its worst" that a patient rates from 0-10 (0 meaning no sweating at all, and 10 meaning worst possible sweating). This single score was used from the number of responses listed below while patient was on active drug, and while they were on placebo. Patients completed this questionnaire daily throughout the study (4 weeks of glycopyrronium cloths, 1 week of washout, and 4 weeks of placebo). Therefore, each patient could have up to 28 entries, however, some patients ended the study early, and some missed a few surveys.
Time Frame: 4 weeks
Population: Patients completed this questionnaire daily throughout the study (4 weeks of active drug, 1 week washout, 4 weeks of placebo).
Measure: Mean (Standard Deviation); unit: score on a scale of 0-10
Units Other Than Participants: Each survey response score
Groups:
- Glycopyrronium Cloths: Patients who received glycopyrronium cloths (either in the first 4 weeks or last 4 weeks of the study).
- Placebo: Participants that received placebo cloths either in the first 4 weeks or last 4 weeks of the study.
Arm/Group | Glycopyrronium Cloths | Placebo
Number analyzed (Participants) | 13 | 13
Number analyzed (Each survey response score) | 210 | 198
score on a scale of 0-10 | 1.2 (2.0) | 3.6 (2.9)

ADVERSE EVENTS:
Time Frame: 17 months
Groups:
- Glycopyrronium Cloths: Participants Randomized to glycopyrronium cloths.
  glycopyrronium cloths: Qbrexza is an anticholinergic indicated for topical treatment of axillary hyperhidrosis in adults and pediatric patients 9 years of age and older
- Placebo: Participants that are randomized to placebo cloths.
  Placebo: Placebo for this study are cloths that look like the qbrexza cloths but do not have any active ingredient.
Arm/Group | Glycopyrronium Cloths | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/13
Other Adverse Events (participants affected / at risk) | 5/13 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrronium Cloths (N=13) | Placebo (N=13)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient could not empty bladder
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrronium Cloths (N=13) | Placebo (N=13)
Dry Mouth (General disorders) | 2 (2) | 0 (0) — Dry Mouth
Folliculitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — Inflammation of hair follicles
Anhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Not sweating systemically
Exacerbated asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Worsening of asthma
Irritant contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — rash due to skin irritant
cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cyst on skin
vertigo (Nervous system disorders) | 0 (0) | 1 (1) — Dizziness
generalized fatigue (General disorders) | 0 (0) | 1 (1) — Tiredness
Lupus Flare (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Flare of lupus

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT04924036/Prot_SAP_000.pdf